CLINICAL TRIAL: NCT01924351
Title: A Phase II Study of Stereotactic Radiosurgery Plus HER-2 Directed Therapy in HER2-positive Breast Cancer With Brain Metastasis
Brief Title: HER2-positive Breast Cancer With Brain Metastasis (GCC 1345)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00056720
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer With Brain Metastasis
Keywords: Breast Cancer with Brain Metastasis; HER2-positive; HER-2 therapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HER2-positive Breast Cancer with Brain Metastasis (Other): Stereotactic Radiosurgery plus HER-2 directed therapy in HER2-positive Breast Cancer with Brain Metastasis
  Interventions: Radiation: Stereotactic Radiosurgery plus HER-2 directed therapy in HER2-positive Breast Cancer with Brain Metastasis

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery plus HER-2 directed therapy in HER2-positive Breast Cancer with Brain Metastasis

SUMMARY:
Primary Objective:

To determine if treatment with SRS followed by a HER-2 directed therapy regimen results in a 6-month distant brain relapse rate of less than 30%.

Secondary Objectives:

1. Describe the natural history of neurocognitive function for women with brain metastases treated with SRS and HER-2 directed systemic therapy and establish a reference benchmark to generate hypothesis for future design of a phase III trial.
2. Describe patterns of distant brain relapse after SRS for all patients and compare them between (a) patients with 1-3 vs. 4-10 brain metastasis and (b) between patients treated with each systemic therapy regimen
3. Describe patterns of neurologic death
4. Describe patterns of local brain relapse
5. Describe patterns of re-irradiation with WBRT or SRS
6. Describe adverse events

DETAILED DESCRIPTION:
Metastatic breast cancer is a leading cause of death for women. HER2(human epidermal growth factor receptor type 2)-positive disease represents a more aggressive type of breast cancer which often afflicts younger patients. As many as one-third of patients with HER2-positive breast cancer develop brain metastasis[1]. The development of brain metastasis in this young female population is particularly devastating as they are often highly functional and may have young children. Improvement in quality of life by preventing neurocognitive decline from disease progression and/or treatment related side effects is paramount.

Patients with 1-10 brain metastasis from HER2+ breast cancer, after informed consent, will be treated with:

Radiosurgery: Gamma-knife, Cyberknife, or linac-based SRS is followed by anti-HER2 based systemic therapy, with the treatment selection of approved agents at the physician's discretion. Possible anti-HER2 agents include trastuzumab, pertuzumab, trastuzumab-emtansine, or lapatinib. Anti-HER2 therapy will be delivered in combination with appropriate cytotoxic therapy as per FDA indications.

Anti-HER2 based systemic therapy will continue until progression, patient discontinuation, unacceptable toxicity or if, in the view of the physician it is no longer indicated.

MRI and neurocognitive testing will be done prior to SRS and repeated every 3 months during the first 6 months from enrollment.

Patients can only be enrolled after all eligibility criteria are met. The date of registration/enrollment is considered to be the day the Eligibility Checklist is signed by the verifying physician. Once a patient is enrolled, a unique case number will be assigned to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis HER2-positive breast cancer. Her2-positive is defined as follows:

  * Validated IHC assay score of 3+ (defined as uniform, intense staining of >30% of invasive tumor cells)
* OR- Average HER2 gene copy number of >6
* OR- Gene amplified (HER2:D17Z1 ratio >2.20).
* Patients with 1-10 newly diagnosed brain metastases
* The contrast-enhancing intraparenchymal brain tumor must be well circumscribed and must have a maximum diameter of ≤ 4.0 cm in any direction on the enhanced scan. If multiple lesions are present and one lesion is at the maximum diameter, the other(s) must not exceed 3.0 cm in maximum diameter.
* History and physical with neurological examination, steroid documentation, height, and weight within 14 days of registration.
* A diagnostic contrast-enhanced MRI of the brain must be performed within 28 days prior to registration.
* Eligibility for treatment with SRS confirmed by a radiation oncologist.
* Performance Status 0-2
* Age ≥ 18.
* CBC with differential obtained within 14 days prior to registration, with adequate bone marrow function defined as follows:
* Absolute neutrophil count (ANC) ≥ 1,100 cells/mm3.
* Platelets ≥ 75,000 cells/mm3.
* Hemoglobin ≥ 9.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥9.0 g/dl is acceptable).
* Adequate renal function within 14 days prior to registration, as defined below:
* BUN ≤ 30 mg/dl.
* Creatinine ≤ 1.5 x ULN
* Creatinine clearance ≥30 mL/min.

Adequate hepatic function within 14 days prior to registration, as defined below:

* Total Bilirubin ≤1.5 x ULN
* ALT/AST ≤ 2.5 x upper limit of normal (ULN).
* Systolic blood pressure ≤ 160 mg Hg or diastolic pressure ≤ 90 mg Hg within 14 days prior to registration.
* Prothrombin time/international normalized ratio (PT INR) < 1.4 for patients not on warfarin confirmed by testing within 14 days prior to registration. Patients on full-dose anticoagulants (e.g., warfarin or LMW heparin) must meet both of the following criteria:
* No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices).
* In-range INR (between 2.5 and 3.5) on a stable dose of warfarin-based oral anticoagulant; or on a stable dose of low molecular weight heparin; or INR between 1.5 and 2 if a Greenfield filter is in place.
* Patient must provide study specific informed consent prior to study entry.
* For women of child-bearing potential, negative serum pregnancy test within 14 days prior to registration.
* Women of childbearing potential and male participants must practice adequate contraception.
* Echocardiogram or MUGA scan with ejection fraction within normal institution limits within 28 days of registration

Exclusion Criteria:

* Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥ 3 years. For example, carcinoma in situ of the oral cavity and cervix are all permissible.
* Leptomeningeal metastases
* Previous treatment with all of the following: lapatinib, trastuzumab, pertuzumab, and trastuzumab emtansine. (Patients are eligible if treated with 3 or less of these agents.)
* Prior cranial radiotherapy.
* Prior resection of cerebral metastases
* Allergy to gadolinium

Severe, active co-morbidity, defined as follows:

* Unstable angina and/or congestive heart failure within the last 6 months.
* Transmural myocardial infarction within the last 6 months.
* New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to registration.
* History of stroke, cerebral vascular accident (CVA) or transient ischemic attack within 6 months.
* Serious and inadequately controlled cardiac arrhythmia.
* Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy.
* Serious or non-healing wound, ulcer, or bone fracture or history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess, major surgical procedure or significant traumatic injury within 28 days prior to registration, with the exception of the craniotomy for tumor resection or follow-on craniotomies to manage complications of brain tumor management such as hemorrhage or infection.
* Bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
* Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration.
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for coagulation parameters are not required for entry into this protocol.
* Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity.
* Any other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy.
* Cognitive impairment that precludes a patient from acting as his or her own agent to provide informed consent.
* Women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the chemotherapeutic treatment involved in this study is potentially teratogenic.
* Pregnant or lactating women, due to possible adverse effects on the developing fetus or infant due to study treatment.
* Patients treated on any other therapeutic clinical protocols within 30 days prior to study entry or during participation in the study.
* Inability to undergo MRI (e.g., due to safety reasons, such as presence of a pacemaker).
* Inability to undergo SRS due to claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Relaspe Rate (Primary) | 12 months
  To determine if treatment with SRS followed by a HER-2 directed therapy regimen results in a 6-month distant brain relapse rate of less than 30%.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Nichols, M.D., Principal Investigator — Univerysity of Maryland Baltimore
Locations (1):
- Ummc Msgcc, Baltimore, Maryland, United States